CLINICAL TRIAL: NCT01895933
Title: The Aim of This Study is to Evaluate the Efficacy and Safety of the Investigational Device, SurgiShield Anti-Adhesion Barrier Gel Made by D Med
Brief Title: Efficacy and Safety of the Investigational Device, SurgiShield Anti-Adhesion Barrier Gel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: D.med (Industry)
Collaborators: Dankook University (Other); Chungbuk National University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DMED-SS001
Record Dates: First submitted 2013-07-08; First posted 2013-07-11 (Estimated); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Wound Healing
Keywords: Investigational device (chitosan gel); Wound healing; Endoscopic sinus surgery; SurgiShield

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active / control (Active Comparator): One side has been treated with SurgiShield
  Interventions: Device: 5ml surgishield
- No intervention (No Intervention): One side has no intervention

INTERVENTIONS:
Device: 5ml surgishield — in the case of active, apply solution type adhesion barrier to merocel and pack 5ml of adhesion inhibitor Surgi Shield on the surgical site
  merocel in the inflated state maintained for 36~48 hours, remove packing then solution type adhesion inhibitor is to be injected in to the surgical site
  Arms: Active / control

SUMMARY:
This clinical trial is intended to evaluate the impact, efficacy, and safety of Chitosan formulated adhesion inhibitor, SurgiShield when used in the process of wound healing after endoscopic sinus surgery.

ELIGIBILITY:
Inclusion Criteria:

* older than 21 years of age
* both side sinusitis
* will undergo endoscopic sinus surgery
* volunteers with informed consent and signature

Exclusion Criteria:

* suppressed immunity patient
* systemic grave condition
* pregnant
* cancer
* severe disease patients
* asthma patients
* AIDS
* cystic fibrosis
* ciliary immobility syndrome
* neutropenia neutrophil
* immunoglobulin deficiency
* wound healing immune disease
* severe liver disease
* severe kidney disease
* lymph or blood clotting disorder or patients treated with coagulants
* patients taking oral or parenteral glucose for diabetes thrombocytopenia
* infectious disease
* currently lactating
* severe septal deviation
* case where there is a severe difference in sinusitis state between sides of nose: there is a 3 or more score difference on the Lund-Mackey CT scan scoring system PNS(ParaNasalSinus)
* shellfish allergy
* food allergy
* had endoscopic sinus surgery in the past
* patient with large sinus polyps
* patients who have received treatment for extrasinus complication

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Adhesion Rate | at 2 weeks
  Adhesion rate at 2 weeks after ESS(endoscopic sinus surgery)

SECONDARY OUTCOMES:
Adhesion Rate | at 1 and 4 weeks
  Adhesion rate at 1 and 4 weeks after ESS(endoscopic sinus surgery) Bleeding score at 0,2,4,6,8,10 minutes after ESS

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Chungbook National University Hospital, Chungju, ChoongChungBukDo
  - Dankook University Hospital, Cheonan, Chungcheongnam-do